CLINICAL TRIAL: NCT04826809
Title: A New Fully-reusable, Affordable, Comfortable Mask Design With Superior Filtration and Fit for Use During Respirator Shortages and Pandemics
Brief Title: New Reusable Mask Design With Superior Filtration and Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Janielle R. Nordell, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-011897
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Covid19; Tuberculosis; Respiratory Viral Infection
Keywords: PPE; mask; N95; pandemic; mask shortage
MeSH Terms: conditions — COVID-19; Tuberculosis | interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Health care workers (Experimental): Health care workers will complete a fit test while wearing the Nordell Single E-100 layer + (cotton layer) mask, Nordell Double E-100 layer mask and an N95 mask
  Interventions: Device: N95 mask; Device: Nordell single E-100 layer mask; Device: Nordell double E-100 layer mask

INTERVENTIONS:
Device: N95 mask — Standard 1870 N95 one time use mask
Device: Nordell single E-100 layer mask — Nordell mask design using one layer of E-100 fabric plus cotton fabric overlay
Device: Nordell double E-100 layer mask — Nordell mask design using two layers of E-100 fabric

SUMMARY:
This study will test the filtration, air leak, and breathability of a newly designed fully washable mask developed by Dr. Nordell with the Mayo Clinic. This mask is theorized to be a superior alternative to other respirators currently used when one-time-use N95 masks are unavailable.

DETAILED DESCRIPTION:
The purpose of this study is to determine potential effectiveness of a new, reusable mask against SARS-CoV-2 and other microbes. This requires filtering down to at least 0.3 microns, as the SARS-CoV-2 virus is on average 0.25-0.5 microns in diameter.

Dr. Nordell has developed a machine-washable mask which shows potential to be significantly more effective than other masks on the market. It uses a fabric that is machine washable, without need for a filter or replaceable component. This fabric, Evolon-100 or E-100, is a microfilament fabric produced by a private company outside of the USA (and is therefore not yet FDA approved as of December 2020).

Unofficial data shows this mask passes the "N95 fit test" before and after multiple washes on the majority of individuals tested, and the material used in Dr. Nordell's design filters 93-96% of 0.3 micron particles. For reference, the N95 mask used in the hospital (whenever concern for potential exposure to COVID-19 or similar contagion exists) filters 95% of 0.3 micron particles when factoring in air leak, assessed with the "fit test." Voluntary survey of users also shows it is more comfortable than other masks, including the N95. This mask is also reported to be breathable even after prolonged use.

This mask design addresses every factor in respirator design. The design intentionally uses pleats to increase the effective mask surface area while decreasing the seal perimeter, resulting in increased air flow, lower pressure drop, and increased filtration efficiency. The investigators propose that it has a higher filtration ability than other washable fabrics tested, filtering at least 93% of 0.3 micron particles, even up to 96%. It also helps prevent air leak, a large factor limiting efficacy of most non-standard masks. It is easy to don and doff, and it is very easy to clean and disinfect. This material can be washed multiple times in a standard washing machine without reducing its effectiveness. And finally, it is very affordable, with materials for one mask costing less than $1.50. All materials used beyond this specific fabric are easily purchased on the internet or in a fabric store.

Upon completion of this research, the investigators hope to demonstrate that this mask is a superior alternative in multiple settings, including hospitals in developing countries with little or no N95 mask access, non-hospital settings such as businesses and schools, as well as for the general population, especially those with high risk for COVID-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Current employee of Mayo Clinic Health System-Mankato
* Passed N95 fit test within the past year
* No medical history of: high blood pressure, current or recent pneumonia or upper respiratory infection, and no uncontrolled chronic asthma
* Ideally with wide representation of genders, race, age, BMI, occupation/role in hospital.
* Willing and able to provde verbal consent.

Exclusion Criteria:

- History of uncontrolled asthma, pneumonia, or hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janielle R Nordell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System in Mankato, Mankato, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Care Workers
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Health Care Workers
Number analyzed (Participants) | 41
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 29 years | 3
  Between 30 and 39 years | 15
  Between 40 and 49 years | 11
  Between 50 and 59 years | 8
  >= 60 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 37
  Hispanic | 2
  Black/African American | 0
  Asian/Pacific Islander | 2
  American Indian | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Fit Tests
Description: Number of participants to pass the respirator fit testing using Bitrix solution. If participants do not smell or taste the solution while wearing the respirator it is considered passed.
Time Frame: Baseline
Population: One participant was excluded from analysis of this outcome measure due to recent viral illness
Measure: Count of Participants; unit: Participants
Groups:
- Health Care Workers: Health care workers will complete a fit test while wearing the Nordell Single E-100 layer + (cotton layer) mask, Nordell Double E-100 layer mask and an N95 mask N95 mask: Standard 1870 N95 one time use mask Nordell single E-100 layer mask: Nordell mask design using one layer of E-100 fabric plus cotton fabric overlay Nordell double E-100 layer mask: Nordell mask design using two layers of E-100 fabric
Arm/Group | Health Care Workers
Number analyzed (Participants) | 40
Participants
  Fit Test N95 | 39
  Fit Test Nordell Single Layer Mask | 39
  Fit Test Nordell Double Layer Mask | 40

2. Primary Outcome: Comfort Level of Nordell Double E-100 Layer Mask
Description: Measured by a self-reported questionnaire that rates the comfort level of the Nordell Double E-100 layer mask on a scale from 0 to 5 (0 is the most uncomfortable mask ever worn, 5 is the best, most comfortable mask)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Health Care Workers
Number analyzed (Participants) | 41
Participants
  0 = most uncomfortable | 0
  1 | 1
  2 | 0
  3 | 4
  4 | 22
  5 = most comfortable | 14

3. Primary Outcome: Ability to Breathe With Nordell Double E-100 Layer Mask
Description: Measured by a self-reported questionnaire that rates ability to breathe comfortably while wearing the Nordell Double E-100 Layer Mask, from 0 (not able to breathe at all) to 5 (just as easy to breathe as not wearing any mask)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Health Care Workers
Number analyzed (Participants) | 41
Participants
  0 (worst) | 0
  1 | 0
  2 | 1
  3 | 4
  4 | 11
  5 (best) | 25

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all subject during participation for approximately 2-3 hours.
Arm/Group | Health Care Workers
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-12-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04826809/Prot_000.pdf